CLINICAL TRIAL: NCT04052997
Title: A Phase 2, Open-Label, Single-Arm Study to Evaluate the Efficacy and Safety of Camidanlumab Tesirine (ADCT-301) in Patients With Relapsed or Refractory Hodgkin Lymphoma
Brief Title: Study to Evaluate the Efficacy and Safety of Camidanlumab Tesirine (ADCT-301) in Patients With Relapsed or Refractory Hodgkin Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ADC Therapeutics S.A. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ADCT-301-201; 2018-002556-32 (EudraCT Number)
Record Dates: First submitted 2019-08-07; First posted 2019-08-12 (Actual); Results first posted 2024-03-28 (Actual); Last update posted 2024-03-28 (Actual); Status verified 2024-03

CONDITIONS: Relapsed Hodgkin Lymphoma; Refractory Hodgkin Lymphoma
Keywords: Camidanlumab Tesirine; Relapsed or Refractory Hodgkins Lymphoma; Classical Hodgkins Lymphoma; Lymphoma
MeSH Terms: conditions — Hodgkin Disease; Recurrence; Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Camidanlumab Tesirine (Experimental): Camidanlumab Tesirine is administered as a 30- minute intravenous (IV) infusion on Day 1 of each cycle (every 3 weeks). Camidanlumab Tesirine will be administered at a dose of 45 μg/kg every 3 weeks for 2 cycles, then 30 μg/kg for subsequent cycles.
  Interventions: Drug: Camidanlumab Tesirine

INTERVENTIONS:
Drug: Camidanlumab Tesirine — Intravenous Infusion
  Other Names: ADCT-301

SUMMARY:
The purpose of this study is to evaluate the clinical efficacy and safety of Camidanlumab Tesirine (ADCT-301) in participants with relapsed or refractory Hodgkin Lymphoma (HL).

DETAILED DESCRIPTION:
This is a phase 2, multi-center, open-label, single-arm study of efficacy and safety of Camidanlumab Tesirine (ADCT-301) in participants with relapsed or refractory Hodgkin lymphoma. This study will enroll approximately 100 participants.

Camidanlumab Tesirine (ADCT-301) is an antibody drug conjugate (ADC), composed of the human monoclonal antibody, HuMax®-TAC, which is directed against human CD25. The antibody is conjugated through a protease cleavable linker to SG3199, a pyrrolobenzodiazepine (PBD) dimer cytotoxin.

For each participant the study will include a screening period (of up to 28 days), a treatment period (cycles of 3 weeks), and a follow-up period (approximately every 12-week visits) for up to 3 years after treatment discontinuation.

Participants may continue treatment for up to 1 year or until disease progression, unacceptable toxicity, or other discontinuation criteria, whichever occurs first.

Additionally, patients benefiting clinically at 1 year may continue treatment after a case by case review with the Sponsor.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent must be obtained prior to any procedures.
2. Male or female participant aged 18 years or older. (16 years or older at US based sites)
3. Pathologic diagnosis of classical Hodgkin lymphoma (cHL).
4. Patients with relapsed or refractory cHL, who have received at least 3 prior lines of systemic therapy (or at least 2 prior lines in HSCT ineligible patients) including brentuximab vedotin and a checkpoint inhibitor approved for cHL (e.g., nivolumab or pembrolizumab). Note 1: Receipt of HSCT to be included in the number of prior therapies needed to meet eligibility.
5. Measurable disease as defined by the 2014 Lugano Classification.
6. Availability of formalin-fixed paraffin-embedded (FFPE) tumor tissue block (or minimum 10 freshly cut unstained slides if block is not available).

   Note 1: Any biopsy since initial diagnosis is acceptable, but if several samples are available, the most recent sample is preferred.

   Note 2: If a sufficient amount of tissue is not available, a fresh biopsy may be taken, provided the procedure is not deemed high-risk and is clinically feasible, and provided it is approved locally.
7. Eastern Cooperative Oncology Group (ECOG) performance status 0-2.
8. Adequate organ function as defined by Screening laboratory values within the following parameters:

   1. Absolute neutrophil count (ANC) ≥ 1.0 × 103/μL (off growth factors at least 72 h).
   2. Platelet count ≥ 75 × 103/μL without transfusion in the past 2 weeks.
   3. ALT, AST, or GGT ≤ 2.5 × the upper limit of normal (ULN) if there is no liver involvement; ALT or AST ≤ 5 × ULN if there is liver involvement.
   4. Total bilirubin ≤ 1.5 × ULN (participants with known Gilbert's syndrome may have a total bilirubin up to ≤ 3 × ULN with direct bilirubin ≤ 1.5 × ULN).
   5. Blood creatinine ≤ 3.0 × ULN or calculated creatinine clearance ≥ 30 mL/min by the Cockcroft-Gault equation.

   Note: A laboratory assessment may be repeated a maximum of two times during the Screening Period to confirm eligibility.
9. Negative beta-human chorionic gonadotropin (β-HCG) pregnancy test within 7 days prior to start of study drug for women of childbearing potential.
10. Women of childbearing potential (WOCBP) must agree to use a highly effective method of contraception from the time of giving informed consent until at least 9.5 months after the last dose of Camidanlumab Tesirine. Men with female partners who are of childbearing potential must agree to use a highly effective method of contraception from the time of giving informed consent until at least 6.5 months after the participants receives his last dose of Camidanlumab Tesirine.

Exclusion Criteria:

1. Previous treatment with Camidanlumab Tesirine.
2. Participation in another investigational interventional study. Being in follow-up of another investigational study is allowed.
3. Known history of hypersensitivity to or positive serum human anti-drug antibody (ADA) to a CD25 antibody.
4. Allogenic or autologous transplant within 60 days prior to start of study drug.
5. Active graft-versus-host disease (GVHD), except for non-neurologic symptoms as a manifestation of mild (≤ Grade 1) chronic GVHD.
6. Post-transplantation lymphoproliferative disorders.
7. Active second primary malignancy other than non-melanoma skin cancers, non-metastatic prostate cancer, in situ cervical cancer, ductal or lobular carcinoma in situ of the breast, or other malignancy that the Sponsor's medical monitor and Investigator agree and document should not be exclusionary.
8. History of symptomatic autoimmune disease (e.g., rheumatoid arthritis, systemic progressive sclerosis [scleroderma], systemic lupus erythematosus, Sjögren's syndrome, autoimmune vasculitis [e.g., Wegener's granulomatosis]) (subjects with vitiligo, type 1 diabetes mellitus, residual hypothyroidism, hypophysitis due to autoimmune condition only requiring hormone replacement may be enrolled).
9. History of neuropathy considered of autoimmune origin (e.g., polyradiculopathy including Guillain-Barré syndrome and myasthenia gravis) or other central nervous system autoimmune disease (e.g., poliomyelitis, multiple sclerosis).
10. History of recent infection (within 4 weeks of Cycle 1, Day 1 [C1D1]) considered to be caused by one of the following pathogens: HSV1, HSV2, VZV, EBV, CMV, measles, Influenza A, Zika virus, Chikungunya virus, mycoplasma pneumonia, Campylobacter jejuni, or enterovirus D68, or severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2).

    Note: An influenza test and a pathogendirected SARS CoV-2 test (such as polymerase chain reaction) are mandatory and must be negative before initiating study treatment (tests to be performed 3 days or less prior to dosing on C1D1; an additional 2 days are allowed in the event of logistical issues for receiving the results on time).
11. Participants known to be or having been infected with human immunodeficiency (HIV) virus, hepatitis B virus (HBV), or hepatitis C virus (HCV), and require anti-viral therapy or prophylaxis. Note: Serology testing is mandatory for patients with unknown status.
12. History of Stevens-Johnson syndrome or toxic epidermal necrolysis.
13. Failure to recover ≤ Grade 1 (Common Terminology Criteria for Adverse Events version 4.0 [CTCAE v4.0]) from acute non-hematologic toxicity (except ≤ Grade 2 neuropathy or alopecia), due to previous therapy, prior to screening.
14. Hodgkin lymphoma (HL) with central nervous system involvement, including leptomeningeal disease.
15. Clinically significant third space fluid accumulation (i.e., ascites requiring drainage or pleural effusion that is either requiring drainage or associated with shortness of breath).
16. Breastfeeding or pregnant.
17. Significant medical comorbidities, including uncontrolled hypertension (blood pressure [BP] ≥ 160/100 mmHg repeatedly), unstable angina, congestive heart failure (greater than New York Heart Association class II), electrocardiographic evidence of acute ischemia, coronary angioplasty or myocardial infarction within 3 months prior to screening, severe uncontrolled atrial or ventricular cardiac arrhythmia, poorly controlled diabetes, or severe chronic pulmonary disease.
18. Major surgery, radiotherapy, chemotherapy, or other anti-neoplastic therapy, within 14 days prior to start of study drug, except shorter if approved by the Sponsor.
19. Use of any other experimental medication within 30 days prior to start of study drug.
20. Any live vaccine within 4 weeks prior to start of study drug and planned live vaccine administration after starting study drug.
21. Congenital long QT (measure between Q wave and T wave in the electrocardiogram) syndrome, or a corrected QTc interval of ≥ 480 ms, at screening (unless secondary to pacemaker or bundle branch block).
22. Any other significant medical illness, abnormality, or condition that would, in the Investigator's judgment, make the participants inappropriate for study participation or put the participant at risk.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 117 (Actual)
Dates: Start 2019-09-13 (Actual); Primary Completion 2023-01-19 (Actual); Study Completion 2023-01-19 (Actual)

CONTACTS AND LOCATIONS:
Locations (73):
- United States (24):
  - Mayo Clinic - Arizona, Scottsdale, Arizona
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - UCSF Health - Hematology and Blood and Marrow Transplant Clinic, San Francisco, California
  - Stanford University Medical Center, Stanford, California
  - Baptist MD Anderson Cancer Center, Jacksonville, Florida
  - Mayo Clinic - Jacksonville, Jacksonville, Florida
  - Northside Hospital - Atlanta, Atlanta, Georgia
  - The University of Chicago Medicine, Chicago, Illinois
  - Norton Cancer Institute - Saint Matthews, Louisville, Kentucky
  - University of Minnesota, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Washington University School of Medicine in Saint Louis, St Louis, Missouri
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Memorial Sloan-Kettering Cancer Center - New York, New York, New York
  - Stony Brook University Cancer Center, Stony Brook, New York
  - University Hospitals Seidman Cancer Center, Cleveland, Ohio
  - Cleveland Clinic - Taussig Cancer Center, Cleveland, Ohio
  - The Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Hollings Cancer Center, Charleston, South Carolina
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - The University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Virginia Cancer Specialists, Fairfax, Virginia
  - Froedtert Hospital, Milwaukee, Wisconsin
- Belgium (5):
  - Algemeen Ziekenhuis Sint-Jan Brugge-Oostende - Campus Sint-Jan, Bruges
  - Cliniques Universitaires Saint-Luc, Brussels
  - Grand Hôpital de Charleroi - Notre Dame, Charleroi
  - Hôpital de Jolimont, La Louvière
  - Centre Hospitalier Universitaire Universite Catholique de Louvain - Site Godinne, Yvoir
- Canada (3):
  - British Columbia Cancer Agency, Vancouver, British Columbia
  - The Ottawa Hospital - General Campus, Ottawa
  - Princess Margaret Cancer Centre, Toronto
- Czechia (3):
  - Fakultní Nemocnice Brno, Brno
  - Fakultní Nemocnice Královské Vinohrady, Prague
  - Vseobecna fakultni nemocnice v Praze, Prague
- France (8):
  - Hôpitaux Universitaires Henri Mondor, Créteil
  - Hôpital François Mitterrand, Dijon
  - Clinique Victor Hugo Le Mans, Le Mans
  - Hôpital Saint-Eloi, Montpellier
  - Hôpital Haut-Lévêque, Pessac
  - Centre Hospitalier Lyon-Sud, Pierre-Bénite
  - Hôpital Pontchaillou, Rennes
  - Centre de Lutte Contre le Cancer - Centre Henri-Becquerel, Rouen
- Universitätsklinikum Halle, Halle, Germany
- Hungary (2):
  - Debreceni Egyetem Klinikai Központ, Debrecen
  - Pécsi Tudományegyetem, Pécs
- Italy (5):
  - Azienda Ospedaliera Nazionale SS. Antonio e Biagio e C. Arrigo - Alessandria, Alessandria
  - Azienda Ospedaliero-Universitaria di Bologna Policlinico Sant Orsola-Malpighi, Bologna
  - Istituto Clinico Humanitas, Milan
  - Istituto Nazionale Tumori IRCCS Fondazione G. Pascale, Napoli
  - Istituto Oncologico Veneto - IRCCS, Padua
- Poland (2):
  - Szpital Wojewódzki w Opolu, Opole
  - Dolnośląskie Centrum Transplantacji Komórkowych z Krajowym Bankiem Dawców Szpiku, Wroclaw
- Spain (14):
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Universitari Vall d'Hebrón, Barcelona
  - Hospital Clínic de Barcelona, Barcelona
  - Institut Català d'Oncologia - Hospital Duran i Reynals (ICO L'Hospitalet), Barcelona
  - Hospital General Universitario Gregorio Marañón, Madrid
  - Hospital Universitario Fundación Jiménez Díaz, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario HM Sanchinarro, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital Universitario Quirónsalud Madrid, Pozuelo de Alarcón
  - Complejo Asistencial Universitario de Salamanca - Hospital Clínico, Salamanca
  - Hospital Clínico Universitario de Valencia, Valencia
  - Hospital Universitari i Politècnic La Fe, Valencia
- United Kingdom (6):
  - NHS Greater Glasgow and Clyde, Glasgow
  - University College London Hospitals NHS Foundation Trust, London
  - The Royal Marsden NHS Foundation Trust, London
  - The Christie NHS Foundation Trust, Manchester
  - Oxford University Hospitals NHS Foundation Trust, Oxford
  - University Hospitals Plymouth NHS Trust, Plymouth

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Herrera AF, Ansell SM, Zinzani PL, Radford J, Maddocks K, Pinto A, Collins GP, Bachanova V, Bartlett NL, Bence-Bruckler I, Hamadani M, Kline J, Mayer J, Savage KJ, Advani RH, Caimi PF, Casasnovas RO, Feldman T, Hess B, Bastos-Oreiro M, Iyengar S, Szomor A, Townsend W, Andre M, Dyczkowski J, Havenith K, Toukam M, Pantano S, Cruz HG, Wang L, Negievich Y, Lucero M, Wuerthner J, Carlo-Stella C. Camidanlumab tesirine for relapsed or refractory classic Hodgkin lymphoma: a phase 2 study. Blood Adv. 2025 Dec 9;9(23):6205-6217. doi: 10.1182/bloodadvances.2024015600. PMID 40811783

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled from September 2019 to January 2023 across 9 countries (USA, Canada, Belgium, Czech Republic, France, Hungary, Italy, Spain, UK).
Pre-assignment Details: Participants with relapsed or refractory Hodgkin Lymphoma received intravenous (IV) infusions of camidanlumab tesirine.
Groups:
- Camidanlumab Tesirine: Participants received IV infusions of camidanlumab tesirine every 3 weeks (Q3W) at a dose of 45 µg/kg on Day 1 of each cycle (one cycle = 21 days) for 2 cycles, followed by 30 µg/kg for subsequent cycles.
Period: Overall Study
Arm/Group | Camidanlumab Tesirine
Started | 117
Discontinued From Study | 117
Completed | 1
Not Completed | 116
Not completed — Withdrawal by Subject | 17
Not completed — Physician Decision | 50
Not completed — Death | 43
Not completed — Lost to Follow-up | 5
Not completed — Progression of Disease | 1

BASELINE CHARACTERISTICS:
Population: All-Treated Population: All participants who received at least 1 dose of camidanlumab tesirine. This population was used in the primary analyses of efficacy and safety.
Groups:
- Camidanlumab Tesirine: Participants received IV infusions of camidanlumab tesirine Q3W at a dose of 45 µg/kg on Day 1 of each cycle (one cycle = 21 days) for 2 cycles, followed by 30 µg/kg for subsequent cycles.
Arm/Group | Camidanlumab Tesirine
Number analyzed (Participants) | 117
Age, Continuous [Mean (Standard Deviation); unit: Years] | 42.5 (16.24)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44
  Male | 73
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7
  Not Hispanic or Latino | 104
  Unknown or Not Reported | 6
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 5
  White | 101
  Other | 5
  Missing | 2
Eastern Cooperative Oncology Group (ECOG) Performance Status Score [Count of Participants; unit: Participants] — The ECOG Performance Status is a scale used to assess a person's level of functioning in terms of their ability to care for themselves, daily activity, and physical ability. The scale consists of 6 grades, ranging from 0 to 5. A grade of 0 indicates the person is fully active and able to carry on as normal, and a grade of 5 indicates death.
  Participants
    ECOG Score 0 | 64
    ECOG Score 1 | 47
    ECOG Score 2 | 6
    ECOG Score 3 | 0

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR)
Description: ORR according to the 2014 Lugano classification as determined by central review in all-treated participants.ORR will be defined as the proportion of participants with a best overall response (BOR) of complete response (CR) or partial response (PR). Data from the All-treated Population.
Time Frame: Up to 3 years
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Camidanlumab Tesirine
Number analyzed (Participants) | 117
Participants | 82

2. Secondary Outcome: Duration of Response (DOR)
Description: DOR defined as the time from the first documentation of tumor response to disease progression or death.
Time Frame: Up to 3 years
Population: Data from participants in the All-Treated Population who achieved ether CR or PR by independent reviewer.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Camidanlumab Tesirine
Number analyzed (Participants) | 82
Months | 13.73 [7.85 to 14.65]

3. Secondary Outcome: CR Rate
Description: CR rate defined as the number of treated participants with a best overall response (BOR) of CR.
Time Frame: Up to 3 years
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Camidanlumab Tesirine
Number analyzed (Participants) | 117
Participants | 39

4. Secondary Outcome: Relapse-Free Survival (RFS)
Description: RFS defined as the time from the documentation of CR to disease progression or death.
Time Frame: Up to 3 years
Population: Data from participants in the All-Treated Population who achieved CR.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Camidanlumab Tesirine
Number analyzed (Participants) | 39
Months | 11.07 [7.36 to NA] — Upper confidence interval was not reached due to lack of events.

5. Secondary Outcome: Progression-Free Survival (PFS)
Description: PFS defined as the time from first dose of study drug until the first date of either disease progression or death due to any cause.
Time Frame: Up to 3 years
Population: as for baseline characteristics
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Camidanlumab Tesirine
Number analyzed (Participants) | 117
Months | 9.13 [5.26 to 14.98]

6. Secondary Outcome: Overall Survival (OS)
Description: OS defined as the time from first dose of study drug until death due to any cause.
Time Frame: Up to 3 years
Population: as for baseline characteristics
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Camidanlumab Tesirine
Number analyzed (Participants) | 117
Months | NA [NA to NA] — Median and confidence intervals were not reached due to lack of events.

7. Secondary Outcome: Number of Participants Who Received Hematopoietic Stem Cell Transplant (HSCT)
Description: Participants receiving HSCT following camidanlumab tesirine, and without any other anticancer therapy in between, other than the therapies preparing for HSCT, were included in this analysis.
Time Frame: Up to 3 years
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Camidanlumab Tesirine
Number analyzed (Participants) | 117
Participants | 18

8. Secondary Outcome: Number of Participants Who Experienced At Least One Treatment-Emergent Adverse Event (TEAE)
Description: An adverse event (AE) is defined as any untoward medical occurrence in a participant or clinical investigation where participants are administered a pharmaceutical product, which does not necessarily have to have a causal relationship with this treatment. A TEAE is defined as an AE that occurs or worsens in the period extending from the first dose of study drug to 30 days after the last dose of study drug in this study or start of a new anticancer therapy/procedure, whichever comes earlier. Clinically significant changes in vital signs, clinical laboratory results, and electrocardiogram were reported as AEs.
Time Frame: Up to 3 years
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Camidanlumab Tesirine
Number analyzed (Participants) | 117
Participants | 116

9. Secondary Outcome: Number of Participants Who Experienced At Least One Serious Adverse Event (SAE)
Description: An SAE is defined as any adverse event (AE) that:
  * results in death.
  * is life threatening.
  * requires inpatient hospitalization or prolongation of existing hospitalization (hospitalization for elective procedures or for protocol compliance is not considered an SAE).
  * results in persistent or significant disability/incapacity.
  * is a congenital anomaly/birth defect.
  * important medical events that do not meet the preceding criteria but based on appropriate medical judgement may jeopardize the participant or may require medical or surgical intervention to prevent any of the outcomes listed above. Clinically significant changes in vital signs, clinical laboratory results, and electrocardiogram were reported as AEs.
Time Frame: Up to 3 years
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Camidanlumab Tesirine
Number analyzed (Participants) | 117
Participants | 46

10. Secondary Outcome: Number of Participants With ECOG Performance Status Score of 0-3 at the End of Trial (EOT)
Description: The ECOG Performance Status is a scale used to asses a person's level of functioning in terms of their ability to care for themselves, daily activity, and physical ability. The scale consists of 6 grades, ranging from 0 to 5. A grade of 0 indicates the person is fully active and able to carry on as normal, and a grade of 5 indicates death.
Time Frame: EOT (up to 3 years)
Population: All-Treated Population: All participants who received at least 1 dose of camidanlumab tesirine and reported ECOG data at EOT. This population was used in the primary analyses of efficacy and safety.
Measure: Count of Participants; unit: Participants
Arm/Group | Camidanlumab Tesirine
Number analyzed (Participants) | 96
Participants
  Score 0 | 43
  Score 1 | 37
  Score 2 | 12
  Score 3 | 4

11. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of Camidanlumab Tesirine Total Antibody
Time Frame: Cycle 1 (one cycle = 21 days): day 1 (predose, EOI, 4h postdose), day 8 (168h), day 15 (336h). Cycle 2: day 1 (predose, EOI, 4h postdose), day 8 (168h), day 15 (336h)
Population: PK Population: The analysis only included participants who received study drug and had at least 1 pre-Cycle 1 Day 1 and 1 post-dose valid (measurable) assessment. Due to the nature of the studied drug (antibody-drug conjugate), some PK parameters frequently could not be measured, or could be measured only briefly.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/L
Arm/Group | Camidanlumab Tesirine
Number analyzed (Participants) | 111
µg/L
  Cycle 1 | 825 (66.7)
  Cycle 2: number analyzed (Participants) | 108
  Cycle 2 | 797 (62.3)

12. Secondary Outcome: Cmax of Camidanlumab Tesirine Unconjugated Warhead SG3199
Time Frame: as for outcome 11
Population: as for outcome 11
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/L
Arm/Group | Camidanlumab Tesirine
Number analyzed (Participants) | 8
µg/L
  Cycle 1 | 0.0170 (31.6)
  Cycle 2: number analyzed (Participants) | 4
  Cycle 2 | 0.0180 (38.3)

13. Secondary Outcome: Cmax of Camidanlumab Tesirine PBD-Conjugated Antibody
Time Frame: as for outcome 11
Population: as for outcome 11
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/L
Arm/Group | Camidanlumab Tesirine
Number analyzed (Participants) | 114
µg/L
  Cycle 1 | 696 (66.5)
  Cycle 2: number analyzed (Participants) | 106
  Cycle 2 | 685 (61.7)

14. Secondary Outcome: Area Under the Plasma Concentration-Time Curve From Time 0 to the End of the Dosing Interval (AUCtau) For Camidanlumab Tesirine Total Antibody
Time Frame: Cycle 2 (one cycle = 21 days): day 1 (predose, EOI, 4h postdose), day 8 (168h), day 15 (336h)
Population: as for outcome 11
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: day*ug/L
Arm/Group | Camidanlumab Tesirine
Number analyzed (Participants) | 111
day*ug/L | 4037 (73.2)

15. Secondary Outcome: AUCtau For Camidanlumab Tesirine PBD-Conjugated Antibody
Time Frame: Cycle 2 (one cycle = 21 days): day 1 (predose, EOI, 4h postdose), day 8 (168h), day 15 (336h)
Population: as for outcome 11
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: day*ug/L
Arm/Group | Camidanlumab Tesirine
Number analyzed (Participants) | 114
day*ug/L | 3067 (65.8)

16. Secondary Outcome: AUCtau For Camidanlumab Tesirine Unconjugated Warhead SG3199
Description: No data collected for this endpoint.
Time Frame: Cycle 2 (one cycle = 21 days): day 1 (predose, EOI, 4h postdose), day 8 (168h), day 15 (336h)
Population: No data collected for this endpoint.
Arm/Group | Camidanlumab Tesirine
Number analyzed (Participants) | 0

17. Secondary Outcome: Area Under the Plasma Concentration-Time Curve From Time 0 to the Time of the Last Quantifiable Concentration (AUClast) For Camidanlumab Tesirine Total Antibody
Time Frame: as for outcome 11
Population: as for outcome 11
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: day*ug/L
Arm/Group | Camidanlumab Tesirine
Number analyzed (Participants) | 111
day*ug/L
  Cycle 1 | 489 (788)
  Cycle 2: number analyzed (Participants) | 108
  Cycle 2 | 725 (897)

18. Secondary Outcome: AUClast For Camidanlumab Tesirine PBD-Conjugated Antibody
Time Frame: as for outcome 11
Population: as for outcome 11
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: day*ug/L
Arm/Group | Camidanlumab Tesirine
Number analyzed (Participants) | 114
day*ug/L
  Cycle 1 | 345 (607)
  Cycle 2: number analyzed (Participants) | 106
  Cycle 2 | 497 (824)

19. Secondary Outcome: AUClast For Camidanlumab Tesirine Unconjugated Warhead SG3199
Time Frame: as for outcome 11
Population: as for outcome 11
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: day*ug/L
Arm/Group | Camidanlumab Tesirine
Number analyzed (Participants) | 8
day*ug/L
  Cycle 1 | 0 (104)
  Cycle 2: number analyzed (Participants) | 4
  Cycle 2 | 0 (211)

20. Secondary Outcome: Area Under the Plasma Concentration-Time Curve From Time 0 to Infinity (AUCinf) For Camidanlumab Tesirine Total Antibody
Time Frame: Cycle 1 (one cycle = 21 days): day 1 (predose, EOI, 4h postdose), day 8 (168h), day 15 (336h)
Population: as for outcome 11
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: day*µg/L
Arm/Group | Camidanlumab Tesirine
Number analyzed (Participants) | 2
day*µg/L | 6473 (11.9)

21. Secondary Outcome: AUCinf For Camidanlumab Tesirine PBD-Conjugated Antibody
Time Frame: Cycle 1 (one cycle = 21 days): day 1 (predose, EOI, 4h postdose), day 8 (168h), day 15 (336h)
Population: as for outcome 11
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: day*µg/L
Arm/Group | Camidanlumab Tesirine
Number analyzed (Participants) | 3
day*µg/L | 5478 (31.2)

22. Secondary Outcome: AUCinf For Camidanlumab Tesirine Unconjugated Warhead SG3199
Time Frame: Cycle 1 (one cycle = 21 days): day 1 (predose, EOI, 4h postdose), day 8 (168h), day 15 (336h)
Population: as for outcome 11
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: day*µg/L
Arm/Group | Camidanlumab Tesirine
Number analyzed (Participants) | 8
day*µg/L | NA (NA) — Geometric mean was not quantifiable due to the low level of observations.

23. Secondary Outcome: Clearance (CL) For Camidanlumab Tesirine Total Antibody
Time Frame: Cycle 1 (one cycle = 21 days): day 1 (predose, EOI, 4h postdose), day 8 (168h), day 15 (336h)
Population: as for outcome 11
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/day
Arm/Group | Camidanlumab Tesirine
Number analyzed (Participants) | 2
L/day | 0.556 (47.9)

24. Secondary Outcome: CL For Camidanlumab Tesirine PBD-Conjugated Antibody
Time Frame: Cycle 1 (one cycle = 21 days): day 1 (predose, EOI, 4h postdose), day 8 (168h), day 15 (336h)
Population: as for outcome 11
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/day
Arm/Group | Camidanlumab Tesirine
Number analyzed (Participants) | 3
L/day | 0.733 (34.7)

25. Secondary Outcome: CL For Camidanlumab Tesirine Unconjugated Warhead SG3199
Time Frame: Cycle 1 (one cycle = 21 days): day 1 (predose, EOI, 4h postdose), day 8 (168h), day 15 (336h)
Population: as for outcome 11
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/day
Arm/Group | Camidanlumab Tesirine
Number analyzed (Participants) | 8
L/day | NA (NA) — Geometric mean was not quantifiable due to the low level of observations.

26. Secondary Outcome: Clearance at Steady State (CLss) For Camidanlumab Tesirine Total Antibody
Time Frame: Cycle 2 (one cycle = 21 days): day 1 (predose, EOI, 4h postdose), day 8 (168h), day 15 (336h)
Population: as for outcome 11
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/day
Arm/Group | Camidanlumab Tesirine
Number analyzed (Participants) | 55
L/day | 0.874 (75.6)

27. Secondary Outcome: CLss For Camidanlumab Tesirine PBD-Conjugated Antibody
Time Frame: Cycle 2 (one cycle = 21 days): day 1 (predose, EOI, 4h postdose), day 8 (168h), day 15 (336h)
Population: as for outcome 11
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/day
Arm/Group | Camidanlumab Tesirine
Number analyzed (Participants) | 54
L/day | 0.958 (64.1)

28. Secondary Outcome: CLss For Camidanlumab Tesirine Unconjugated Warhead SG3199
Time Frame: Cycle 2 (one cycle = 21 days): day 1 (predose, EOI, 4h postdose), day 8 (168h), day 15 (336h)
Population: as for outcome 11
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/day
Arm/Group | Camidanlumab Tesirine
Number analyzed (Participants) | 8
L/day | NA (NA) — Geometric mean was not quantifiable due to the low level of observations.

29. Secondary Outcome: Apparent Terminal Elimination Half-Life (T1/2) For Camidanlumab Tesirine Total Antibody
Time Frame: as for outcome 11
Population: as for outcome 11
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: day
Arm/Group | Camidanlumab Tesirine
Number analyzed (Participants) | 6
day
  Cycle 1: number analyzed (Participants) | 2
  Cycle 1 | 5.91 (68.6)
  Cycle 2 | 4.46 (24.6)

30. Secondary Outcome: T1/2 For Camidanlumab Tesirine PBD-Conjugated Antibody
Time Frame: as for outcome 11
Population: as for outcome 11
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: day
Arm/Group | Camidanlumab Tesirine
Number analyzed (Participants) | 6
day
  Cycle 1: number analyzed (Participants) | 3
  Cycle 1 | 3.89 (17.5)
  Cycle 2 | 4.05 (26.1)

31. Secondary Outcome: T1/2 For Camidanlumab Tesirine Unconjugated Warhead SG3199
Time Frame: as for outcome 11
Population: as for outcome 11
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: day
Arm/Group | Camidanlumab Tesirine
Number analyzed (Participants) | 8
day
  Cycle 1 | NA (NA) — Geometric mean was not quantifiable due to the low level of observations.
  Cycle 2 | NA (NA) — Geometric mean was not quantifiable due to the low level of observations.

32. Secondary Outcome: Volume of Distribution at Steady State (Vss) For Camidanlumab Tesirine Total Antibody
Time Frame: as for outcome 11
Population: as for outcome 11
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L
Arm/Group | Camidanlumab Tesirine
Number analyzed (Participants) | 6
L
  Cycle 1: number analyzed (Participants) | 2
  Cycle 1 | 5.91 (68.6)
  Cycle 2 | 3.14 (44.1)

33. Secondary Outcome: Vss For Camidanlumab Tesirine PBD-Conjugated Antibody
Time Frame: as for outcome 11
Population: as for outcome 11
Measure: Geometric Least Squares Mean (Geometric Coefficient of Variation); unit: L
Arm/Group | Camidanlumab Tesirine
Number analyzed (Participants) | 6
L
  Cycle 1: number analyzed (Participants) | 3
  Cycle 1 | 2.81 (24.9)
  Cycle 2 | 3.17 (37.6)

34. Secondary Outcome: Vss For Camidanlumab Tesirine Unconjugated Warhead SG3199
Time Frame: as for outcome 11
Population: as for outcome 11
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L
Arm/Group | Camidanlumab Tesirine
Number analyzed (Participants) | 8
L
  Cycle 1 | NA (NA) — Geometric mean was not quantifiable due to the low level of observations.
  Cycle 2 | NA (NA) — Geometric mean was not quantifiable due to the low level of observations.

35. Secondary Outcome: Accumulation Index (AI) For Camidanlumab Tesirine Total Antibody
Description: AI is the ratio of area under the serum concentration-time curve (AUC) from 0 to 21 days for Cycle 2 divided by AUC from 0 to 21 days for Cycle 1.
Time Frame: Cycle 1 and 2: day 0 to 21
Population: as for outcome 11
Measure: Geometric Least Squares Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Camidanlumab Tesirine
Number analyzed (Participants) | 8
ratio | 1.30 (52.9)

36. Secondary Outcome: AI For Camidanlumab Tesirine PBD-Conjugated Antibody
Description: AI is the ratio of AUC from 0 to 21 days for Cycle 2 divided by AUC from 0 to 21 days for Cycle 1.
Time Frame: Cycle 1 and 2: day 0 to 21
Population: as for outcome 11
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Camidanlumab Tesirine
Number analyzed (Participants) | 6
ratio | 1.04 (4.00)

37. Secondary Outcome: AI For Camidanlumab Tesirine Unconjugated Warhead SG3199
Description: AI is the ratio of AUC from 0 to 21 days for Cycle 2 divided by AUC from 0 to 21 days for Cycle 1.
Time Frame: Cycle 1 and 2: day 0 to 21
Population: as for outcome 11
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Camidanlumab Tesirine
Number analyzed (Participants) | 8
ratio | NA (NA) — Geometric mean was not quantifiable due to the low level of observations.

38. Secondary Outcome: Number of Participants With Confirmed Positive Anti-Drug Antibody (ADA) Responses Post Dose
Description: Detection of ADAs was performed by using a screening assay for identification of antibody positive samples/participants, a confirmation assay, and titer assessment.
Time Frame: Up to 3 years
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Camidanlumab Tesirine
Number analyzed (Participants) | 117
Participants | 2

39. Secondary Outcome: Change From Baseline in Health-Related Quality of Life (HRQoL) as Measured by EuroQoL-5 Dimensions-5 Levels (EQ-5D-5L) Visual Analog Scale (VAS)
Description: Participants were asked to indicate their health state on a VAS with scores ranging from 'the worst health you can imagine' (score 0) to 'the best health you can imagine' (score 100). Participants are asked to mark an "X" on the VAS to indicate their own health and then to report the score in a text box. Positive changes from Baseline represent an an improvement in heath.
Time Frame: Baseline, Day 1 of Cycles 2 to 15 (one cycle = 21 days) and EOT (up to 3 years)
Population: Patient Reported Outcome (PRO) Population: All participants in the all-treated population with baseline score (at least one instrument) and at least 1 post-baseline score (in at least one instrument).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Camidanlumab Tesirine
Number analyzed (Participants) | 116
score on a scale
  Cycle 2: number analyzed (Participants) | 111
  Cycle 2 | 3.6 (14.41)
  Cycle 3: number analyzed (Participants) | 90
  Cycle 3 | 5.2 (15.14)
  Cycle 4: number analyzed (Participants) | 74
  Cycle 4 | 4.9 (17.65)
  Cycle 5: number analyzed (Participants) | 62
  Cycle 5 | 4.6 (19.66)
  Cycle 6: number analyzed (Participants) | 44
  Cycle 6 | -1.2 (14.97)
  Cycle 7: number analyzed (Participants) | 32
  Cycle 7 | 4.5 (11.88)
  Cycle 8: number analyzed (Participants) | 19
  Cycle 8 | 4.5 (13.24)
  Cycle 9: number analyzed (Participants) | 17
  Cycle 9 | 3.3 (13.74)
  Cycle 10: number analyzed (Participants) | 11
  Cycle 10 | 1.3 (7.30)
  Cycle 11: number analyzed (Participants) | 7
  Cycle 11 | -0.6 (10.44)
  Cycle 12: number analyzed (Participants) | 6
  Cycle 12 | -4.8 (5.31)
  Cycle 13: number analyzed (Participants) | 3
  Cycle 13 | -1.7 (2.89)
  Cycle 14: number analyzed (Participants) | 3
  Cycle 14 | -1.7 (10.41)
  Cycle 15: number analyzed (Participants) | 3
  Cycle 15 | -3.3 (7.64)
  EOT: number analyzed (Participants) | 80
  EOT | -3.1 (20.06)

40. Secondary Outcome: Change From Baseline in HRQoL as Measured by Functional Assessment of Cancer Therapy - Lymphoma (FACT-Lym)
Description: The FACT-Lym consists of a 27-item general core questionnaire (i.e., Functional Assessment of Cancer Therapy - General [FACT-G]) and a 15-item disease-specific questionnaire (Lymphoma Subscale). The FACT-G includes 4 domains: physical well-being, social/family well-being, emotional well-being, and functional well-being. The total FACT-Lym score (0-168) was obtained by summing individual subscale scores. Higher scores for the scales indicate better quality of life. Change was calculated as the value at the last observation minus the value at baseline.
Time Frame: Baseline, Day 1 of Cycles 2 to 15 (one cycle = 21 days) and EOT (up to 3 years)
Population: PRO Population: All participants in the all-treated population with baseline score (at least one instrument) and at least 1 post-baseline score (in at least one instrument).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Camidanlumab Tesirine
Number analyzed (Participants) | 116
score on a scale
  Cycle 2: number analyzed (Participants) | 108
  Cycle 2 | -0.45 (4.079)
  Cycle 3: number analyzed (Participants) | 89
  Cycle 3 | -0.02 (4.935)
  Cycle 4: number analyzed (Participants) | 73
  Cycle 4 | -0.20 (5.384)
  Cycle 5: number analyzed (Participants) | 57
  Cycle 5 | -0.13 (4.906)
  Cycle 6: number analyzed (Participants) | 42
  Cycle 6 | -1.29 (4.318)
  Cycle 7: number analyzed (Participants) | 30
  Cycle 7 | 0.39 (3.892)
  Cycle 8: number analyzed (Participants) | 19
  Cycle 8 | 0.40 (4.419)
  Cycle 9: number analyzed (Participants) | 17
  Cycle 9 | -1.38 (6.262)
  Cycle 10: number analyzed (Participants) | 10
  Cycle 10 | 1.16 (2.374)
  Cycle 11: number analyzed (Participants) | 6
  Cycle 11 | 1.50 (5.167)
  Cycle 12: number analyzed (Participants) | 5
  Cycle 12 | -1.40 (0.548)
  Cycle 13: number analyzed (Participants) | 2
  Cycle 13 | 0.00 (0.000)
  Cycle 14: number analyzed (Participants) | 2
  Cycle 14 | 0.00 (0.000)
  Cycle 15: number analyzed (Participants) | 2
  Cycle 15 | 0.00 (0.000)
  EOT: number analyzed (Participants) | 77
  EOT | -3.06 (6.802)

ADVERSE EVENTS:
Time Frame: Up to 3 years
Description: All AEs, AESIs, and SAEs regardless of relationship to study drug were reported from the time a participant signed the ICF until 30 days after the last dose of study drug. After 30 days following the last dose of study drug, only related SAEs were reported.
Arm/Group | Camidanlumab Tesirine
All-Cause Mortality (participants affected / at risk) | 43/117
Serious Adverse Events (participants affected / at risk) | 46/117
Other Adverse Events (participants affected / at risk) | 116/117
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Camidanlumab Tesirine (N=117)
Bone marrow failure (Blood and lymphatic system disorders) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 1 (1)
Cardiac arrest (Cardiac disorders) | 1 (1)
Left ventricular failure (Cardiac disorders) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1)
Thyroiditis (Endocrine disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 2 (2)
Duodenal ulcer (Gastrointestinal disorders) | 1 (1)
Duodenal ulcer perforation (Gastrointestinal disorders) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (2)
Pyrexia (General disorders) | 3 (3)
Drug-induced liver injury (Hepatobiliary disorders) | 1 (1)
Cellulitis (Infections and infestations) | 2 (2)
Pneumonia (Infections and infestations) | 2 (2)
Adenovirus infection (Infections and infestations) | 1 (1)
Bronchopulmonary aspergillosis (Infections and infestations) | 1 (1)
JC virus infection (Infections and infestations) | 1 (1)
Lung infection (Infections and infestations) | 1 (1)
Pneumonia bacterial (Infections and infestations) | 1 (1)
Pneumonia pneumococcal (Infections and infestations) | 1 (1)
Rash pustular (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Septic shock (Infections and infestations) | 1 (1)
Tooth infection (Infections and infestations) | 1 (1)
Varicella zoster virus infection (Infections and infestations) | 1 (1)
Transplant failure (Injury, poisoning and procedural complications) | 1 (1)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 2 (2)
Acidosis (Metabolism and nutrition disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1)
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Myositis (Musculoskeletal and connective tissue disorders) | 1 (1)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Guillain-Barre syndrome (Nervous system disorders) | 4 (4)
Epilepsy (Nervous system disorders) | 1 (1)
Peripheral motor neuropathy (Nervous system disorders) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1)
Radiculopathy (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Device occlusion (Product Issues) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Tubulointerstitial nephritis (Renal and urinary disorders) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 (3)
Dermatitis exfoliative generalised (Skin and subcutaneous tissue disorders) | 1 (1)
Dermatosis (Skin and subcutaneous tissue disorders) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1)
Lichenoid keratosis (Skin and subcutaneous tissue disorders) | 1 (1)
Parakeratosis (Skin and subcutaneous tissue disorders) | 1 (1)
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 1 (1)
Shock haemorrhagic (Vascular disorders) | 1 (1)
Superior vena cava occlusion (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Camidanlumab Tesirine (N=117)
Anaemia (Blood and lymphatic system disorders) | 29 (39)
Thrombocytopenia (Blood and lymphatic system disorders) | 24 (34)
Neutropenia (Blood and lymphatic system disorders) | 19 (29)
Lymphopenia (Blood and lymphatic system disorders) | 18 (26)
Sinus tachycardia (Cardiac disorders) | 8 (8)
Hypothyroidism (Endocrine disorders) | 12 (12)
Hyperthyroidism (Endocrine disorders) | 8 (8)
Thyroiditis (Endocrine disorders) | 7 (7)
Nausea (Gastrointestinal disorders) | 32 (40)
Constipation (Gastrointestinal disorders) | 20 (23)
Diarrhoea (Gastrointestinal disorders) | 19 (26)
Vomiting (Gastrointestinal disorders) | 13 (17)
Abdominal pain (Gastrointestinal disorders) | 12 (14)
Dry mouth (Gastrointestinal disorders) | 7 (7)
Dyspepsia (Gastrointestinal disorders) | 6 (6)
Stomatitis (Gastrointestinal disorders) | 6 (6)
Fatigue (General disorders) | 45 (53)
Pyrexia (General disorders) | 35 (47)
Oedema peripheral (General disorders) | 14 (15)
Chills (General disorders) | 12 (14)
Asthenia (General disorders) | 8 (8)
Face oedema (General disorders) | 7 (7)
Upper respiratory tract infection (Infections and infestations) | 7 (8)
Gamma-glutamyltransferase increased (Investigations) | 20 (26)
Alanine aminotransferase increased (Investigations) | 15 (16)
Aspartate aminotransferase increased (Investigations) | 14 (17)
Blood alkaline phosphatase increased (Investigations) | 11 (15)
Amylase increased (Investigations) | 9 (12)
Lipase increased (Investigations) | 9 (11)
Weight decreased (Investigations) | 9 (9)
Hypophosphataemia (Metabolism and nutrition disorders) | 21 (29)
Hyperglycaemia (Metabolism and nutrition disorders) | 14 (21)
Hypokalaemia (Metabolism and nutrition disorders) | 14 (18)
Decreased appetite (Metabolism and nutrition disorders) | 12 (12)
Hypomagnesaemia (Metabolism and nutrition disorders) | 9 (10)
Hyponatraemia (Metabolism and nutrition disorders) | 7 (9)
Dehydration (Metabolism and nutrition disorders) | 6 (7)
Arthralgia (Musculoskeletal and connective tissue disorders) | 19 (22)
Myalgia (Musculoskeletal and connective tissue disorders) | 11 (15)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6 (9)
Headache (Nervous system disorders) | 19 (22)
Dizziness (Nervous system disorders) | 12 (13)
Peripheral sensory neuropathy (Nervous system disorders) | 7 (7)
Dysgeusia (Nervous system disorders) | 6 (6)
Neuropathy peripheral (Nervous system disorders) | 6 (6)
Insomnia (Psychiatric disorders) | 16 (17)
Anxiety (Psychiatric disorders) | 6 (8)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 16 (18)
Cough (Respiratory, thoracic and mediastinal disorders) | 12 (12)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 10 (11)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 38
Rash (Skin and subcutaneous tissue disorders) | 31 (36)
Pruritus (Skin and subcutaneous tissue disorders) | 28 (30)
Erythema (Skin and subcutaneous tissue disorders) | 14 (19)
Dry skin (Skin and subcutaneous tissue disorders) | 7 (8)
Hypertension (Vascular disorders) | 6 (9)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2022-02-16): https://cdn.clinicaltrials.gov/large-docs/97/NCT04052997/Prot_000.pdf
  • Statistical Analysis Plan (2022-09-13): https://cdn.clinicaltrials.gov/large-docs/97/NCT04052997/SAP_001.pdf